CLINICAL TRIAL: NCT04656080
Title: AlloSure Test Characteristics in Immunologically Quiescent and Immunologically Active Heart Transplant Recipients: Does Maximal Cardiopulmonary Stress Testing Prior to Assay Preserve Test Specificity While Enhancing Sensitivity?
Brief Title: Cardiopulmonary Stress Testing (CPET) AlloSure Study
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 020-188
Record Dates: First submitted 2020-10-06; First posted 2020-12-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Transplant; Failure, Heart
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transplant recipients <1year without AMR: 20 recent transplant recipients (<1 year) without antibody-mediated rejection (AMR);
  Interventions: Behavioral: CPET exercise testing
- 3 months post-heart transplant with AMR: • 7 transplant recipients, at least 3 months post-transplant, with antibody-mediated rejection
  Interventions: Behavioral: CPET exercise testing

INTERVENTIONS:
Behavioral: CPET exercise testing — * The cardiopulmonary exercise testing (CPET) is done.
  * EKG testing will be done as part of the CPET test. Allosure testing will be done at baseline and then at 1 hr, 4 hrs, 1 day, 7 days after CPET.

SUMMARY:
1. Cell-free DNA does not vary significantly as a function of the activity of immunologically quiescent cardiac transplant recipients, despite the metabolic demands of the transplanted organ. (The implication of the null result would be that no restrictions to patient activity, nor modification of cardiac rehabilitation prescription, would be necessary to maintain proper test characteristics of AlloSure testing).
2. In immunologically active cardiac transplant allografts, exercise prior to assay of donor-derived cell-free DNA can be used to increase the sensitivity of the AlloSure test. (The implication of this would be that the optimal time-frame for drawing an Allosure may actually be post-exercise, and that window will be characterized).

DETAILED DESCRIPTION:
The specific research questioned aimed to be addressed with this proposed study are:

i. Are dd-cfDNA levels in heart transplant recipients independent of recent cardiopulmonary exercise? More specifically, does the metabolic demand of maximal cardiopulmonary exercise in recent heart transplant recipients trigger a release of dd-cfDNA (if so, then what is the time course for resolution back to baseline?) ii. If dd-cfDNA does not release to any significant degree with cardiac allografts with short donor-ischemic time, does this test characteristic continue to hold for cardiac allografts transplanted after longer donor ischemic times? iii. In cardiac transplant recipients with medically stabilized, treated antibody-mediated rejection (AMR) and persistent dd-cfDNA elevation, does a discrete episode of maximal cardiometabolic activity trigger any additional elevation of dd-cfDNA, and again, with what time course?

ELIGIBILITY:
Inclusion Criteria:

Post-orthotopic heart transplant patients

Exclusion Criteria:

1. orthopedic, neurologic and/or any other limitations that do not allow for exercise testing on a treadmill or cycle ergometer;
2. individuals who require supplemental oxygen or have current permanent tracheostomies will be excluded from this study;
3. individuals who are discharged to a long-term acute care facility;
4. skilled nursing facility or with palliative care or hospice care will be excluded; (e) inmates and pregnant women;

(f) patients with antibody-mediate rejection that are not felt to be safe for cardiopulmonary stress testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects to be enrolled in this study will be male and/or female hemodynamically stable outpatients who have undergone orthotopic heart transplant within three months from enrollment date for the recent transplant cohort, and within 10 years of transplant for the antibody-mediated rejection cohort. All subjects will be 18 to 80 years of age. All subjects must be able to read and understand an informed consent to be enrolled in the study.
  For the stabilized antibody-mediated rejection cohort, only patients with invasive coronary angiography indicating no more than ISHLT grade 1 coronary allograft vasculopathy within 6 months prior to testing will be included.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
• Cell-free DNA (AlloSure) levels after maximal cardiopulmonary exercise | 10 days
  • Cell-free DNA (AlloSure) levels after maximal cardiopulmonary exercise
• Comparison of maximal oxygen consumption (VO2) | 10 days
  • Comparison of maximal oxygen consumption (VO2)
• Comparison of level of cell-free DNA | 10 days
  Comparison of level of cell-free DNA

SECONDARY OUTCOMES:
• Time-dependent changes in high-sensitivity troponin-levels | 10 days
  • Time-dependent changes in high-sensitivity troponin-levels

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gottlieb, MD, Principal Investigator — BSWRI
Locations (1):
- Baylor Scott & White health research institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Snyder MW, Kircher M, Hill AJ, Daza RM, Shendure J. Cell-free DNA Comprises an In Vivo Nucleosome Footprint that Informs Its Tissues-Of-Origin. Cell. 2016 Jan 14;164(1-2):57-68. doi: 10.1016/j.cell.2015.11.050. PMID 26771485